CLINICAL TRIAL: NCT01813526
Title: Evaluation of an Elemental Formula in Infants With Protein Sensitive Colitis
Brief Title: Infants With Protein Sensitive Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: AH75
Record Dates: First submitted 2013-03-14; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Protein Sensitive Colitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Infant Formula (Experimental): Experimental formula to be fed ad libitum.
  Interventions: Other: Experimental Infant Formula

INTERVENTIONS:
Other: Experimental Infant Formula — Nutritionally complete free amino acid-based medical food.
  Other Names: EleCare

SUMMARY:
Infants with protein sensitive colitis fed a nutritionally complete free amino acid-based medical food will be evaluated for 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 6 months of age
* 36-42 weeks gestational age at birth
* Singleton or Twin birth
* Diagnosed with protein sensitive colitis
* Negative stool culture at time of study entry
* No previous history of consuming free amino acid-based medical food
* Not receiving cisapride or steroids
* No vitamin mineral supplement administration during the study period with the exception of iron or fluoride
* No milk or soy products for the duration of the study

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 1999-11; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Physician Rated Symptom Score | Study Day (SD) 1 and 43
  Calculated from a symptom checklist based on parent report of the previous 7 day history; Change in physician rated symptom score from SD 1 to SD 43.

SECONDARY OUTCOMES:
Mean Rank Stool Consistency | Study Day (SD) 2-4 and 40-42
  Parent reported stool records
Weight | Study Day (SD) 1 and 43 Visits
  Weight gain during the feeding period
Formula Intake | Study Day (SD) 2-4 and 40-42
  Parent reported records of formula intake
Daily Stool Number | Study Day (SD) 2-4 and 40-42
  Parent reported stool records
Stool Occult Blood | Study Day (SD) 2-4 and 40-42
  Parent collected sample of infant stool

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, RD, Study Chair
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital, Omaha, Nebraska

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765